CLINICAL TRIAL: NCT03368391
Title: Pulpal Blood Flow With the Use of Intra-nasal Anesthetic: a Randomized Double-blind Crossover Study
Brief Title: : Pulpal Blood Flow With the Use of Intra-nasal Anesthetic
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Janice Townsend, Associate Professor, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 9924
Record Dates: First submitted 2017-11-30; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Local Anesthetic Drug Adverse Reaction; Local Infiltration; Pulp Disease, Dental
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Tetracaine; Oxymetazoline; Lidocaine; Epinephrine; Mepivacaine

STUDY DESIGN:
Intervention Model Description: triple blinded cross over randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: the dentist who administered the study medications will know their identity but the participant, investigator who tests the teeth, and person calling for later outcomes will not know.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Sequence 1 (Other): All participants will be exposed to all study medications during 3 subsequent visits with a 1 week washout between visits.
  Sequence 1 participants will receive the drugs in the following sequence: 1) tetracaine HCl and oxymetazoline HCl 2) 3% mepivacaine 3) 2% lidocaine with 1:100,000 epi
  Interventions: Drug: tetracaine HCl and oxymetazoline HCL; Drug: 2% Lidocaine with 1:100,000 epinephrine; Drug: 3% Mepivacaine with 1:100,000 epinephrine; Drug: saline intranasal; Drug: saline infiltration
- Sequence 2 (Other): All participants will be exposed to all study medications during 3 subsequent visits with a 1 week washout between visits.
  Sequence 2 participant will receive the drugs in the following sequence: 1) 2% lidocaine with 1:100,000 epi 2) tetracaine HCl and oxymetazoline HCl 3) 3% mepivacaine
  Interventions: Drug: tetracaine HCl and oxymetazoline HCL; Drug: 2% Lidocaine with 1:100,000 epinephrine; Drug: 3% Mepivacaine with 1:100,000 epinephrine; Drug: saline intranasal; Drug: saline infiltration
- Sequence 3 (Other): All participants will be exposed to all study medications during 3 subsequent visits with a 1 week washout between visits.
  Sequence 3 participants will receive the drugs in the following sequence: 1) 3% mepivacaine 2) 2% lidocaine with 1:100,000 epi 3) tetracaine HCl and oxymetazoline HCl
  Interventions: Drug: tetracaine HCl and oxymetazoline HCL; Drug: 2% Lidocaine with 1:100,000 epinephrine; Drug: 3% Mepivacaine with 1:100,000 epinephrine; Drug: saline intranasal; Drug: saline infiltration

INTERVENTIONS:
Drug: tetracaine HCl and oxymetazoline HCL — 0.4 mL HCl and oxymetazoline HCl administered intranasally
Drug: 2% Lidocaine with 1:100,000 epinephrine — 2.5 mL of 2% Lidocaine with 1:100,000 epi will be infiltrated at anterior teeth
Drug: 3% Mepivacaine with 1:100,000 epinephrine — 2.5 mL of 3% Mepivacaine will be infiltrated at anterior teeth
Drug: saline intranasal — 0.4 mL intranasal saline will be administered as a placebo
Drug: saline infiltration — 2.8 mL of saline will be infiltrated at anterior teeth as a placebo

SUMMARY:
Anesthetics with vasoconstrictors decrease pulpal blood flow but the impact of intranasal local anesthetics on blood flow is unknown. This blinded, randomized crossover clinical trial will compare the effects of different local anesthetics on anterior teeth in healthy volunteers. On separate study visits patients will receive either traditional injections or intranasal administration of the following solutions: 2% lidocaine with 1:100,000 epi, 3% mepivacaine, tetracaine HCl and oxymetazoline HCl, or saline. The following variables will be assessed: pulpal blood flow, pulpal sensibility, pain on administration, and adverse outcomes.

DETAILED DESCRIPTION:
Informed Consent Prior to screening, informed consent will be obtained from subjects by study personnel. All questions pertaining to the study will be addressed and answered prior to the participants' agreement to voluntarily partake. The informed consent explicitly states that participation, failure to participate, or withdrawal from the study will not impact the employment or educational standing or any student or employee.

Participants who are screened, selected, provided informed consent, and partake in the 6-week study will be compensated for their time commitment will receive a total of $100.00. They will receive $25 for the screening/impression visit if accepted and $25 for each of the additional 3 sessions.

Study Medications

2% Lidocaine with 1:100,000 epinephrine is the most commonly used local anesthetic in dentistry. It is associated in with a very small increase in blood pressure and heart rate due to the vasoconstrictor which is clinically insignificant in healthy adults. Reports of true allergy in the literature are very rare in a drug that has been administered millions a times a year for decades. This drug is associated with transient blood flow reduction to the pulp which is inconsequential to a healthy dental pulp but may have an impact on a tooth that has sustained dental injury.

3% mepivacaine is another commonly used local anesthetic. It has less inherent vasodilating properties than other local anesthetics and can be used without a vasoconstrictor. This drug has been shown to have a reduced impact on pulpal blood flow. However, 3% mepivacaine has a much shorter duration of action due to the lack of vasoconstrictor and may be of inadequate duration to manage a dental trauma.

Kovanaze is an intranasal local anesthetic that has been FDA approved for use. It is comprised of the local anesthetic tetracaine HCl and oxymetazoline which is the primary ingredient in the drug Afrin. It has been approved for children over 40 kg and adults of all ages. The impact of Kovanaze is unknown but it would be expected to have no impact on blood flow as it is administered in an area distant from the blood vessels that supply teeth.

Saline will be administered as a placebo at each study visit so participants only receive one study drug per session. It will be administered either intranasally or as an injection as the protocol dictates.

Kovanaze® dose syringes will be stored according to manufacturer's label in refrigeration. Injectable anesthetics, in vials, will be stored according to manufacturer's labels. All disposals will comply with manufacturer's labels and meet requirements of those laid out by federal and state regulations. All three drugs are FDA approved for anesthesia of anterior teeth. No drug is contraindicated under any procedural circumstance including trauma at this time and can each be interpreted as fulfilling the standard of care for local anesthesia to manage a traumatic injury.

Group Assignment

Subjects accepted into the study will be randomized into three different groups that will determine the order medications are administered using a random number generator. All groups will be exposed to all three study medications distributed over 3 sessions. Each subject will serve as their own control. There will be a minimum of a one week washout period between study visits.

Clinical Visits

At each clinical visit, participants will receive a 3.0ml buccal infiltration of anesthetic (lidocaine or mepivicaine) or placebo, 0.5ml palatal infiltration of anesthetic (lidocaine or mepivicaine) or placebo, and 0.4ml (2 sprays, 0.4ml of Kovanaze) or saline placebo in right nostril. Buccal and palatal infiltrations will be administered by same operator over a one minute time period. Buccal infiltrations will be administered in labial vestibule above apices of teeth #7 and #8. Palatal infiltration will be administered in attached keratinized gingiva near apices of teeth #7 and #8. Each anesthetic syringe will be labeled accordingly to correspond to material used. The dentist that gives the medicine will know which medicine is being given but the dentist that later tests the teeth will not know so that bias is avoided.

i. First visit Study Groups Testing dosage Placebo Group 1 Kovanaze® (2 sprays in right nostril per manufacture instructions, 0.4ml) Saline buccal infiltrations and palatal infiltration (3.5ml) Group 2 2% lidocaine with 1: 100, 000 epinephrine buccal infiltration and palatal infiltration (3.5ml) Saline nasal dosage in right nostril (0.4ml) Group 3 3% mepivicaine buccal infiltrations and palatal infiltration (3.5ml) Saline nasal dosage in right nostril (0.4ml)

ii. Second visit Study Groups Testing dosage Placebo Group 1 3% mepivicaine buccal infiltrations and palatal infiltration (3.5ml) Saline nasal dosage in right nostril (0.4ml) Group 2 Kovanaze® (2 sprays in right nostril per manufacture instructions, 0.4ml) Saline buccal infiltrations and palatal infiltration (3.5ml) Group 3 2% lidocaine with 1: 100, 000 epinephrine buccal infiltration and palatal infiltration (3.5ml) Saline nasal dosage in right nostril (0.4ml)

iii. Third visit Study Groups Testing dosage Placebo Group 1 2% lidocaine with 1: 100, 000 epinephrine buccal infiltration and palatal infiltration (3.5ml) Saline nasal dosage in right nostril (0.4ml) Group 2 3% mepivicaine buccal infiltrations and palatal infiltration (3.5ml) Saline nasal dosage in right nostril (0.4ml) Group 3 Kovanaze® (2 sprays in right nostril per manufacture instructions, 0.4ml) Saline buccal infiltrations and palatal infiltration (3.5ml)

Individual Sensor Holder

The primary determinant of blood flow will be measured by use of noninvasive, objective laser doppler flowmetry. In order to ensure the laser sensor tip is placed on the same location at each visit a custom holder from dental putty will be fabricated. This is a standard procedure in dentistry and involves placing a malleable material on the teeth. This material sets to a rubbery consistency in a matter of minutes and will allow the study team to adapt the holder for both the laser doppler tip as well as the pulp tester tip.

The pulp tester is a simple instrument, commonly used in daily practice to measure pulp sensitivity. See further explanation below. The screening appointment and fabrication of the sensor holder should not take more than 45 minutes.

Baseline Data Gathering

Prior to any intervention baseline data will be gathered from each patient. An objective measure of blood flow to the teeth with be gathered by noninvasive laser doppler flowmetry which requires placement of a probe on the front of the tooth with the assistance of the custom fabricated holder. Doppler is emerging as the gold standard for assessing pulpal blood flow in research but its exorbitant expense prohibits its widespread use in clinical practice.

The efficacy and duration of the local anesthesia will be subjectively tested through Electric Pulp Testing or EPT. Electric pulp testing tests the sensibility of dental nerves to an electric current and is one of the most commonly used pulp testing modalities due to its lack of harm to the dental pulp, reasonable cost, widespread availability, and acceptability by patients. Every 4 seconds a slight increase in electricity is added until the subject can feel the electricity. Once any sensation is perceived, testing is discontinued and this value is recorded. Patients hold the testing probe to provide grounding and they are told to let go of the probe when they feel sensation precluding any further sensation. This avoids the risk of injury or pain associated with electric pulp testing.

For both of these procedures a plastic, non-latex rubber dam or barrier is placed to prevent interference from the gingiva.

Testing visit

Each testing visit is expected to last no more than 1.5 hours. Participants will be asked to lay in supine position for 10 minutes prior to initiation of testing. To obtund the sensation associated with an injection, 20% benzocaine topical 3min prior to delivery of anesthesia as is the standard in clinical dentistry and trauma management. 2.5 mL of 2% Lidocaine with 1:100,000 epi and 3% Mepivacaine by injection. 0.4 mL of Kovanaze will be administered intranasally.

Laser Doppler Flowmetry readings will be taken at 7, 12, 17, 32, 47, and 62 minutes after administration of anesthetics. Electronic Pulp Testing will be performed at 5, 10, 15, 30, 45, and 60 minutes.

Subjective data, pertaining to pain and comfort with procedure, will be collected using questionnaire. Following delivery of anesthetic or placebo a Heft-Parker Visual Analogue Scale will be utilized to assess pain associated with injection and nasal spray. Patients will be monitored for adverse reactions during the clinical procedure and although rare, most adverse reactions related to local anesthesia are acute. The testing visits should last no more than 90 minutes each.

Upon discharge patients will be reminded to call the emergency contact and seek emergency medical care for major adverse events. This is unexpected as no major adverse events have been recorded with Kovanaze and are not encountered in daily use of lidocaine or mepivacaine. Participants will also be given the take home questionnaire and asked to deliver it to the student researcher. The following will be addressed in the take home questionnaire: Heft-Parker Visual Analogue Scale for pain (1 hour after, 4 hours after, 24 hours after), minor adverse events, and a Likert response scale of patient satisfaction. The questionnaire takes 5 minutes to take for a total of 15 minutes of questionnaire for each testing visit.

Adverse events will be reported to the IRB, LSUHSC, and the Louisiana State Board of Dentistry as required by statute. Compensation for injuries will not be provided by study personnel if an adverse reaction has occurred. Participants will be asked to provide a contact in case of emergency prior to commencement of testing.

Data collected and interpreted from the research study will be only available to those who are a part of the research team. Participants information that is collected during the project will be kept confidential. Participants will be designated a identification number, rather than name. Only the principal investigator and research member designated to the current study will be able to obtain the information gathered by participants identification number. After testing, data collection, documentation of results, and manuscript formulation, all information, including participant identification number, will be safely locked in filing cabinet and/or stored on an encrypted password protected computer, in a secure location.

Data Analysis:

The difference between baseline and experimental values for doppler flowmetry and EPT will be determined and analyzed for each study medication. The means and standard deviations will be plotted and used in statistical measurements for significance. Data will be analyzed using ANOVA and Tukey's method for group comparisons.

Outcomes for the Heft Parker Visual Analogue Scale for pain and the Likert Scale for patient satisfaction will be analyzed using Wilcoxon Rank Sum tests. Reports of adverse events will be categorized and reported using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2 with no contraindications to the medications in this study
* no restorations on the anterior teeth, no sign of history of dental trauma, and a normal periodontium to be included

Exclusion Criteria:

* known hypersensitivity to tetracaine, benzyl alcohol ester local anesthetics, p-aminobenzoic acid (PABA), oxymetazoline, lidocaine, and mepivacaine -inadequately controlled hypertension or thyroid disease, frequent nose bleeds, or history of methemoglobinemia will not be eligible. Patients taking monoamine oxidase inhibitors are not eligible as well. Pregnant women will not be eligible as a precaution.
* Subjects will be excluded if they have restorations, traumatic occlusion, orthodontic appliance, pathologic discoloration of dentition, fixed retainer on maxillary anterior, resorption, pulp canal obliteration, previous endodontic therapy, history of trauma to maxillary anterior dentition, or a fractured tooth structure

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-01-03 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pulpal Blood Flow | baseline and 7, 12, 17, 32, 47, and 62 minutes after administration of anesthetics
  change in pulpal blood flow will be measured using doppler flowmetry

SECONDARY OUTCOMES:
Pulp sensibility | baseline before administration of anesthetics
  pulp sensibility will be measured by a electrical pulp testing unit
Pulp sensibility | 5 minutes after administration of anesthetics
  pulp sensibility will be measured by a electrical pulp testing unit
Pulp sensibility | 10 minutes after administration of anesthetics
  pulp sensibility will be measured by a electrical pulp testing unit
Pulp sensibility | 15 minutes after administration of anesthetics
  pulp sensibility will be measured by a electrical pulp testing unit
Pulp sensibility | 30 minutes after administration of anesthetics
  pulp sensibility will be measured by a electrical pulp testing unit
Pulp sensibility | 45minutes after administration of anesthetics
  pulp sensibility will be measured by a electrical pulp testing unit
Pulp sensibility | 60 minutes after administration of anesthetics
  pulp sensibility will be measured by a electrical pulp testing unit
Pain | baseline before administration of local anesthetics
  pain utilizing Heft Parker Pain Scale
Pain | immediately after administration of local anesthetics
  pain utilizing Heft Parker Pain Scale
Pain | 1 hour after administration of local anesthetics
  pain utilizing Heft Parker Pain Scale
Pain | 4 hours after administration of local anesthetics
  pain utilizing Heft Parker Pain Scale
Pain | 24 hours after administration of local anesthetics
  pain utilizing Heft Parker Pain Scale
adverse outcomes | immediately after administration of local anesthetics
  A list of potential complications will be given to patients and they will check the ones that will apply. This is qualitative not quantitative data so units are not relevant.
Adverse outcomes | 1 hour after administration of local anesthetics
  A list of potential complications will be given to patients and they will check the ones that will apply. This is qualitative not quantitative data so units are not relevant.
Adverse outcomes | 4 hours after administration of local anesthetics
  A list of potential complications will be given to patients and they will check the ones that will apply. This is qualitative not quantitative data so units are not relevant.
Adverse outcomes | 24 hours after administration of local anesthetics
  A list of potential complications will be given to patients and they will check the ones that will apply. This is qualitative not quantitative data so units are not relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Janice A Townsend, DDS, MS, Principal Investigator — LSUHSC School of Dentistry

IPD SHARING:
Plan to Share IPD: No